CLINICAL TRIAL: NCT03533803
Title: Indomethacin Prior to Difficult Embryo Transfer is it a Solution?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Nile Ivf Center, Cairo, Egypt (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Assistant Professor of Obstetrics and Gynaecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12018
Record Dates: First submitted 2018-05-12; First posted 2018-05-23 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Difficult Embryo Transfer
MeSH Terms: interventions — Indomethacin; Suppositories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Indomethacin) (Active Comparator): All patient had long stimulation protocol and IVF/ICSI. After mock embryo transfer women with any degree of difficulty will receive Indomethacin 100Mg Suppository 1-2 hours before embryo transfer.
  Interventions: Drug: Indomethacin 100Mg Suppository; Procedure: IVF/ICSI
- Group B (Control) (Placebo Comparator): All patient had long stimulation protocol and IVF/ICSI. After mock embryo transfer women with any degree of difficulty will not receive any medications before embryo transfer.
  Interventions: Procedure: IVF/ICSI

INTERVENTIONS:
Drug: Indomethacin 100Mg Suppository — Indomethacin 100Mg Suppository will be given 1 to 2 hours before embryo transfer in cases with difficult mock embryo transfer in the active comparator group.
  Other Names: Indomethacin
  Arms: Group A (Indomethacin)
Procedure: IVF/ICSI — patients received induction with the long agonist stimulation protocol. Followed by ovum pickup and embryo transfer. Only those with difficult mock embryo transfer will be recruited in this study.

SUMMARY:
IVF/ICSI patients who had difficult mock embryo transfer on the day of ovum pick up. Will be randomly assigned into two groups; group A will receive 100mg indomethacin rectal suppository 1-2 hours before ET and group B will not receive indomethacin

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients undergoing IVF cycle with difficult mock embryo transfer
* Early follicular FSH level ≤10 IU/L.
* Tubal, male infertility and unexplained causes of fertility will be recruited.
* Fresh ET.

Exclusion Criteria:

* Repeated IVF failure.
* Past history of allergy to NSAID, bronchial asthma , peptic ulcer or inflammatory bowel disease.

  * Easy mock embryo transfer.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 6 weeks
  the number of total gestational sacs divided by the total number of embryos transferred.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 weeks
  Presence of fetal pulsations after 2 weeks from the positive pregnancy test.
Ongoing pregnancy rate | 12 weeks
  Pregnancies continuing beyond 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sarwat Ahawany, MD, Study Chair — Cairo University
Locations (1):
- Nile IVF center, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No